CLINICAL TRIAL: NCT05746611
Title: To Conduct a Phase IV Clinical Trial of Recombinant Mycobacterium Tuberculosis Fusion Protein in Community Population Aged 6 Months and Above.
Brief Title: Phase IV Clinical Study of Recombinant Mycobacterium Tuberculosis Fusion Protein
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Anhui Zhifei Longcom Biologic Pharmacy Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: LKM-2022-EC02
Record Dates: First submitted 2023-02-09; First posted 2023-02-28 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Latent Tuberculosis Infection
MeSH Terms: conditions — Latent Tuberculosis | interventions — Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort 1 (Experimental): Recombinant Mycobacterium Tuberculosis Fusion Protein (EC):
  Dosage form: injection. Main ingredients and contents: Recombinant Mycobacterium tuberculosis fusion protein, 0.3ml, 0.5ml, 1.0ml per bottle.
  1. This product is used alone: 0.1ml (5U) of this product is inhaled and injected into the palmar skin of the forearm by the Mondu's method. 2. This product combined with TB-PPD: 0.1ml(5U) of this product and 0.1ml(5U) of TB-PPD were inhaled respectively, and the product was injected intradermally into the volar side of the left forearm by the Mondu's method. After observing no abnormality for 5 minutes, TB-PPD was injected intradermally into the volar side of the right forearm.
  Purified protein derivative (TB-PPD) :
  Dosage form: Injection. Main components and contents: Purified protein derivative of tuberculin 50IU/ml. 0.1ml (5U) of the product was inhaled and injected into the palmar skin of the forearm by the Mondu's method.
  Interventions: Biological: Recombinant Mycobacterium tuberculosis fusion protein for injection; Biological: TB-PPD was injected
- Cohort 2 (Experimental): Recombinant Mycobacterium Tuberculosis Fusion Protein (EC):
  Dosage form: injection. Main ingredients and contents: Recombinant Mycobacterium tuberculosis fusion protein, 0.3ml, 0.5ml, 1.0ml per bottle.
  1. This product is used alone: 0.1ml (5U) of this product is inhaled and injected into the palmar skin of the forearm by the Mondu's method. 2. This product combined with TB-PPD: 0.1ml(5U) of this product and 0.1ml(5U) of TB-PPD were inhaled respectively, and the product was injected intradermally into the volar side of the left forearm by the Mondu's method. After observing no abnormality for 5 minutes, TB-PPD was injected intradermally into the volar side of the right forearm.
  Interventions: Biological: Recombinant Mycobacterium tuberculosis fusion protein for injection

INTERVENTIONS:
Biological: Recombinant Mycobacterium tuberculosis fusion protein for injection — For the suction test, EC0.1ml was injected into the palmar skin of the forearm by the Mondu's method
Biological: TB-PPD was injected — For the aspiration test, 0.1ml TB-PPD was injected into the palmar skin of the forearm by the Mondu's method
  Arms: Cohort 1

SUMMARY:
Cohort 1 was a randomized, double-blind, controlled clinical trial with a planned enrollment of 500 patients. Cohort 2 is a non-randomized, open-label clinical trial with a planned enrollment of approximately 60000 patients. Cohort I was injected with EC and TB-PPD in both arms, and cohort II was injected with EC only

DETAILED DESCRIPTION:
Assessment of effectiveness:

In cohort 1, the injection site reaction was examined at 0min, 24h, 48h and 72h after skin test, and the transverse and longitudinal diameters of the erythema and induration were measured and recorded in millimeters (mm), the larger the erythema or induration. Any blisters, necrosis, lymphangitis should be faithfully recorded.

In cohort 2, the injection site reaction was examined at 0min and 48-72 h after skin test, and the transverse and longitudinal diameters of the erythema and induration were measured and recorded in millimeters (mm), the larger the erythema or induration. Any blisters, necrosis, lymphangitis should be faithfully recorded.

Safety assessments:

The safety assessment included all expected and unexpected medical events that occurred during the observation period of the clinical trial (within 72 hours after the skin test) and were related or unrelated to the injection of the investigational drug. These included specific reactions such as redness, induration, blister, necrosis, and lymphangitis at the injection site (palmar forearm). Common and occasional adverse reactions include:

Local adverse reactions: injection site pruritus, injection site pain, injection site rash;

Systemic adverse reactions included fever, headache, nausea, fatigue, myalgia, diarrhea, vomiting, paresthesia.

ELIGIBILITY:
Inclusion Criteria:

* People aged 6 months and above (≥6 months).
* Normal armpit body temperature (body temperature below 37.5℃ from 6 months to 14 years old, body temperature below 37.3℃ from 15 years old and above).
* I or my guardian agree to participate in this study and sign the informed consent, willing and able to comply with the requirements of this clinical study protocol.

Exclusion Criteria:

* Patients with acute infectious diseases (such as measles, pertussis, influenza, pneumonia, etc.), acute eye conjunctivitis, acute otitis media, extensive skin diseases and allergic diseases
* A pure protein derivative or similar product was used within 3 months prior to the initiation of this trial.
* Participated in other new drug clinical trials within 3 months prior to clinical trials.
* Any circumstances were considered by the investigators to have the potential to influence the assessment of the trial.

Min Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 7500 (Actual)
Dates: Start 2023-04-17 (Actual); Primary Completion 2024-05-13 (Actual); Study Completion 2024-05-13 (Actual)

PRIMARY OUTCOMES:
In Cohort 1, the diameter of redness or induration at the reaction site | The skin test was performed at 0 minute after injection.
  In cohort 1, the diameter of redness or induration at the reaction site was measured with a scale at 0 minute after skin testing.
In Cohort 1, the diameter of redness or induration at the reaction site | The skin test was performed at 24 hours after injection.
  In cohort 1, the diameter of redness or induration at the reaction site was measured with a scale at 24 hours after skin testing.
In Cohort 1, the diameter of redness or induration at the reaction site | The skin test was performed at 48 hours after injection.
  In cohort 1, the diameter of redness or induration at the reaction site was measured with a scale at 48 hours after skin testing.
In Cohort 1, the diameter of redness or induration at the reaction site | The skin test was performed at 72 hours after injection.
  In cohort 1, the diameter of redness or induration at the reaction site was measured using a scale at 72 hours after skin testing.
In Cohort 2, the diameter of redness or induration at the reaction site | 0 minute after the skin test
  In cohort 2, the diameter of skin redness or induration at the injection site was measured with a scale at 0 minute after the skin test.
In Cohort 2, the diameter of redness or induration at the reaction site | Within 48 to 72 hours after skin testing
  In cohort 2, the diameter of skin redness or induration at the primary injection site was measured with a scale between 48 and 72 hours after skin testing.
Number of cases in which all adverse events occurred. | The skin test was performed 72 hours after injection.
  Number of cases in which all adverse events occurred within 72 hours after skin testing.
Incidence of SAE | Incidence of SAE within 72 hours after full vaccination
  Incidence of SAE within 72 hours after injection

CONTACTS AND LOCATIONS:
Overall Officials: Yi Mo, Master, Principal Investigator — Guangxi Zhuang Autonomous Region Center for Disease Control and Prevention
Locations (1):
- Guangxi Zhuang Autonomous Region Center for Disease Control and Prevention, Liuchow, Guangxi, China

REFERENCES:
- [Derived] Chen J, Zhao L, Zhou X, Mo Y, Kong L, Ma F, Wu L, Huang D, Yang H, Gong L. Safety and Diagnostic Performance of Recombinant Fusion Protein ESAT6-CPF10 Skin Test in A Large Population: A Phase 4 Clinical Trial. J Infect Dis. 2025 Oct 15;232(4):882-891. doi: 10.1093/infdis/jiaf332. PMID 40560769